CLINICAL TRIAL: NCT06090851
Title: Impact of the Daily Consumption of Herbal Pralines on Parameters of Oral Health in Crew Members of a Naval Ship at Sea - a Randomized Controlled Trial
Brief Title: Herbal Pralines - Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yvonne Jockel-Schneider, Prof.Dr., Wuerzburg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAVNIT_23
Record Dates: First submitted 2023-09-18; First posted 2023-10-19 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Periodontitis; Gingivitis
MeSH Terms: conditions — Periodontitis; Gingivitis | interventions — Nitrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- verum (Active Comparator): pralines containing nitrate 3x day (200mg nitrate per day)
  Interventions: Dietary Supplement: herbal nitrate Pralines with nitrate
- placebo (Placebo Comparator): pralines without nitrate
  Interventions: Dietary Supplement: herbal nitrate Pralines without nitrate

INTERVENTIONS:
Dietary Supplement: herbal nitrate Pralines with nitrate — consumption of herbal pralines with nitrate
  Arms: verum
Dietary Supplement: herbal nitrate Pralines without nitrate — consumption of herbal pralines without nitrate
  Arms: placebo

SUMMARY:
This randomized, double-blinded, placebo-controlled two-arm, parallel group clinical trial is designed to evaluate the impact of the consumption of two herbal pralines containing 200 mg nitrate on clinical signs of gingival inflammation (Bleeding on probing) without an accompanied professional mechanical plaque removal.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years,
* minimum of 20 % of the measure points showing a manifest bleeding after probing,
* no periodontal maintenance therapy within the past 4 months,
* a minimum of 10 remaining natural teeth

Exclusion Criteria:

* history of drug / alcohol abuse,
* systemic intake of antibiotics < 6 months prior to the study period,
* regular use of anti-inflammatory drugs,
* regular use of antibacterial mouthwashes,
* known allergic reactions to any ingredient in the experimental pralines
* mean arterial blood pressure MAD <80mmHg
* known allergies and intolerances to any of the ingredients of the experimental pralines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
bleeding on probing (BoP) | baseline
  observed percentage of probing sites being positive for bleeding on probing
bleeding on probing (BoP) | 14 days
  observed percentage of probing sites being positive for bleeding on probing
bleeding on probing (BoP) | 28 days
  observed percentage of probing sites being positive for bleeding on probing

SECONDARY OUTCOMES:
composition of the oral microbiome (subgingival) | baseline
  microbial samples are taking from the tooth showing the highest number of BoP positive sites
composition of the oral microbiome (subgingival) | day 14
  microbial samples are taking from the tooth showing the highest number of BoP positive sites
composition of the oral microbiome (subgingival) | day 28
  microbial samples are taking from the tooth showing the highest number of BoP positive sites
Plaque Control Record (PCR) according to O´Leary | Baseline
  The percentage of plaque coverage will calculated from the number of plaque-covered surfaces in relation to the number of all examined surfaces per tooth.
Plaque Control Record (PCR) according to O´Leary | Day 14
  The percentage of plaque coverage will calculated from the number of plaque-covered surfaces in relation to the number of all examined surfaces per tooth.
Plaque Control Record (PCR) according to O´Leary | Day 28
  The percentage of plaque coverage will calculated from the number of plaque-covered surfaces in relation to the number of all examined surfaces per tooth.
Gingiva Index (GI) | Baseline
  Gingival Index will be assessed strictly visually on a categorial scale ranging from GI 0 to GI 3 according to the Lobene modification
Gingiva Index (GI) | Day 14
  Gingival Index will be assessed strictly visually on a categorial scale ranging from GI 0 to GI 3 according to the Lobene modification
Gingiva Index (GI) | Day 28
  Gingival Index will be assessed strictly visually on a categorial scale ranging from GI 0 to GI 3 according to the Lobene modification
Pocket probing depth | Baseline
  The probable pocket depth (PPD) in mm will recorded using a PCP-11 Marquis periodontal probe (Hu-Friedy, USA) at six measuring points (mesio-buccal, buccal, disto-buccal, disto-oral, oral, mesio-oral) per tooth
Pocket probing depth | Day 14
  The probable pocket depth (PPD)in mm will recorded using a PCP-11 Marquis periodontal probe (Hu-Friedy, USA) at six measuring points (mesio-buccal, buccal, disto-buccal, disto-oral, oral, mesio-oral) per tooth
Pocket probing depth | Day 28
  The probable pocket depth (PPD) in mm will recorded using a PCP-11 Marquis periodontal probe (Hu-Friedy, USA) at six measuring points (mesio-buccal, buccal, disto-buccal, disto-oral, oral, mesio-oral) per tooth
Periodontal inflamed surface area (PISA) mm2 | Day 28
  PISA will be calculated from Pocket probing depth (PPD) in mm, Gingival Recession (Rec) in mm and BoP
Periodontal inflamed surface area (PISA) | Baseline
  PISA will be calculated from PPD, Rec and BoPPISA willl be calculated from Pocket probing depth (PPD), Gingival Recession (Rec) and BoP
Periodontal inflamed surface area (PISA) | Day 14
  PISA will be calculated from Pocket probing depth (PPD), Gingival Recession (Rec) and BoP
Short-term Sick Leave | baseline
  The number of occasions a study participant consulted the onboard physician due to respiratory or gastrointestinal discomfort is documented via a questionnaire. Diagnoses reported by the study participants will be verified by the onboard physician
Short-term Sick Leave | Day 14
  The number of occasions a study participant consulted the onboard physician due to respiratory or gastrointestinal discomfort is documented via a questionnaire. Diagnoses reported by the study participants will be verified by the onboard physician
Short-term Sick Leave | Day 28
  The number of occasions a study participant consulted the onboard physician due to respiratory or gastrointestinal discomfort is documented via a questionnaire. Diagnoses reported by the study participants will be verified by the onboard physician
Salivary nitrate levels | Baseline
  Salivary nitrate levels will be determined from the salivary samples by High-Performance Anion-Exchange Chromatography with Suppressed Conductivity Detection (HPAEC-CD).
Salivary nitrate levels | Day 14
  Salivary nitrate levels will be determined from the salivary samples by High-Performance Anion-Exchange Chromatography with Suppressed Conductivity Detection (HPAEC-CD).
Salivary nitrate levels | Day 28
  Salivary nitrate levels will be determined from the salivary samples by High-Performance Anion-Exchange Chromatography with Suppressed Conductivity Detection (HPAEC-CD).
Salivary nitrite levels | Baseline
  Salivary nitrite levels will be determined from the salivary samples by High-Performance Anion-Exchange Chromatography with Suppressed Conductivity Detection (HPAEC-CD).
Salivary nitrite levels | Day 14
  Salivary nitrite levels will be determined from the salivary samples by High-Performance Anion-Exchange Chromatography with Suppressed Conductivity Detection (HPAEC-CD).
Salivary nitrite levels | Day 28
  Salivary nitrite levels will be determined from the salivary samples by High-Performance Anion-Exchange Chromatography with Suppressed Conductivity Detection (HPAEC-CD).
saliva buffer capacity ( the ability of a buffer solution to resist a change in pH) | baseline
  buffer capacity will be assed by PHmeter datenloGGer-store
saliva buffer capacity ( the ability of a buffer solution to resist a change in pH) | day14
  buffer capacity will be assed by PHmeter datenloGGer-store
saliva buffer capacity ( the ability of a buffer solution to resist a change in pH) | day28
  buffer capacity will be assed by PHmeter datenloGGer-store
saliva PH levels | baseline
  PH levels will be assed by PHmeter datenloGGer-store
saliva PH levels | Day 14
  PH levels will be assed by PHmeter (PHM 230 S) datenloGGer-store
saliva PH levels | Day 28
  PH levels will be assed by PHmeter (PHM 230 S) datenloGGer-store
Bacteria relevant to caries in saliva | Baseline
  Bacteria relevant to caries are cultivated and counted
Bacteria relevant to caries in saliva | Day 14
  Bacteria relevant to caries are cultivated and counted
Bacteria relevant to caries in saliva | Day 28
  Bacteria relevant to caries are cultivated and counted

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - German Naval Medical Institute, Kronshagen
  - Section of Periodontology, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided